CLINICAL TRIAL: NCT01084265
Title: Clinical Trial on Application of Injectable Recombinant Human Luteinizing Hormone (Luveris®) in the Treatment of Chinese Female Patients With Hypogonadotropic Hypogonadism: A Multi-center, Open, Prospective Drug Clinical Trial for Registration
Brief Title: A Study Using Recombinant Human Luteinizing Hormone (r-hLH, Luveris®) in the Treatment of Chinese Women With Hypogonadotropic Hypogonadism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Pte. Ltd., Singapore (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMP25345
Record Dates: First submitted 2010-03-04; First posted 2010-03-10 (Estimated); Results first posted 2012-05-22 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Hypogonadism
Keywords: Hypogonadism; Recombinant human follicle stimulating hormone (r-hFSH); Recombinant leutinizing hormone (r-hLH)
MeSH Terms: conditions — Hypogonadism | interventions — Luteinizing Hormone, beta Subunit; Glycoprotein Hormones, alpha Subunit; follitropin alfa; Chorionic Gonadotropin

INTERVENTIONS:
Drug: Recombinant human luteinizing hormone (r-hLH) — One r-hLH (75 International Units [IU]) injection s.c. once daily.
  Other Names: Luveris (r-hLH)
Drug: Recombinant human follicle-stimulating hormone (r-hFSH) — One r-hFSH (150 IU) injection s.c. once daily.
  Other Names: Gonal-F (r-hFSH)
Drug: Human chorionic gonadotropin (hCG) — After adequate follicular response, ovulation induction was triggered by an injection of 10,000 IU hCG.

SUMMARY:
This was a prospective, open, non-comparative study to evaluate the safety and efficacy of recombinant human luteinizing hormone (rhLH, Luveris) administered subcutaneously (s.c.) in follicular development during ovulation induction in 31 Chinese female subjects with hypogonadotropic hypogonadism.

DETAILED DESCRIPTION:
The objective of this prospective, open, non-comparative study was to assess the safety and efficacy of rhLH (Luveris) administered subcutaneously in follicular development during ovulation induction in Chinese female subjects with hypogonadotropic hypogonadism. The study was organized on an outpatient basis involving a single cycle of treatment. Prior to entry into the study, the diagnosis of hypogonadotropic hypogonadism was confirmed by history, by the presence or absence of specific clinical features and by measuring serum gonadotropin levels. Once a subject has signed the informed consent form and after satisfying all eligibility criteria, the subject received a combination of daily injection of recombinant human follicle-stimulating hormone (rhFSH) 150 international units (IU) plus rhLH 75 IU. After adequate follicular response, ovulation induction was triggered by an injection of 10,000 IU human chorionic gonadotropin (hCG). Luteal phase function was assessed by serum progesterone level determination.

ELIGIBILITY:
Inclusion Criteria:

* Be premenopausal, between 18 and 39 years of age
* Have a clinical history of hypogonadotropic hypogonadism, and laboratory test result comply with diagnosis of hypogonadotropic hypogonadism during screening procedure
* Have discontinued gonadotropins, gonadotropin-releasing hormone (GnRH) (gonadotropin naïve), or estrogen progesterone replacement therapy at least one month before the screening procedure
* Have a negative progestin challenge test performed during screening
* Have the following hormonal values in a centrally analyzed fasting blood sample, drawn within 6 months before initiation of treatment:
* Follicular stimulating hormone (FSH): < 5 international units/liter (IU/L)
* Luteinizing hormone (LH): < 1.2 IU/L
* Oestradiol (E2): < 60 picogram/milliliter (pg/mL) (<220 picomolar/liter [pmol/L])
* Prolactin (PRL): < 44.3 nanogram/milliliter (ng/mL) (< 1040 milli-international units/liter [mIU/L])
* Thyrotrophin-stimulating hormone (TSH): < 6.5 micro-international units (uIU/mL)
* Free Thyroxine (T4): 0.8-1.8 nanogram/deciliter (ng/dL) (11-24 pmol/L)
* Triiodothyronine (T3): < 1.0 ng/mL (< 3.5 nanomolar/liter [nmol/L])
* Have an endovaginal pelvic ultrasound scan showing (i) no ovarian tumor and cyst < 2 centimeters (cm); (ii) no clinically significant uterine abnormality, and (iii) < 13 mm small follicles (mean diameter < 10 mm) on the largest section through each ovary
* Have a normal cervical pap smear within 6 months of the initial visit
* Have a body mass index (BMI) between 18.4 and 31.4 kilogram/meter square (kg/m^2)
* Be willing and able to comply with the protocol for the duration of the study
* Have given written informed consent prior to any study related procedure

Exclusion Criteria:

* Ongoing pregnancy
* Any chronic systemic disease
* Hypersensitive to study drug and control drug
* History of severe ovarian hyperstimulation syndrome
* Abnormal gynecological bleeding of undetermined origin
* Previous or current hormone dependent tumor
* Known active substance abuse or eating disorder
* Known central nervous system (CNS) lesions: In cases where hypogonadotropic hypogonadism (HH) is secondary to a CNS lesion or its treatment, the subject will not be eligible without consulting Serono's Medical Director
* Exercise program exceeding 10 hours per week
* Currently undergoing treatment with psychotropic medication or with any other medication known to interfere with normal reproductive function (for example, neuroleptics, dopamine antagonists)
* There is any abnormality, decided by investigators, which might produce effect on the absorption, distribution and excretion of investigational drug

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2004-02; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xin Li, Study Director — Merck Pte. Ltd., Singapore
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Recombinant Human Luteinizing Hormone (Luveris): Recombinant human luteinizing hormone (rhLH, Luveris) injection 75 international units (IU) subcutaneously (s.c.) daily along with 150 IU recombinant human follicle-stimulating hormone (rhFSH, Gonal-F) s.c. daily for no longer than 14 days unless the diameter of ovarian follicles indicated the maturation (greater than 14 millimeter [mm]).
Period: Overall Study
Arm/Group | Recombinant Human Luteinizing Hormone (Luveris)
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Recombinant Human Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — Demographic data for only "N = 30" participants was reported as 1 participant did not meet the inclusion criteria.
  years | 30.1 (4.09)
Sex: Female, Male [Count of Participants; unit: Participants] — Demographic data for only "N = 30" participants was reported as 1 participant did not meet the inclusion criteria.
  Participants
    Female | 30
    Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Met Both Index 1 and Index 2
Description: The three indices were defined as; Index 1: diameter of at least one follicle is greater than 17 mm; Index 2: serum oestradiol (E2) level in blood serum above 109 picogram/ milliliter (pg/mL) on human chorionic gonadotropin (hCG) injection day; Index 3: participant refuses to take hCG injection for the concern of ovarian hyperstimulation syndrome (OHSS) or participant is pregnant. A subset of these participants met Index 3.
Time Frame: Day 14
Population: Per protocol set included all participants who completely met all the requirements of clinical trial protocol.
Measure: Number; unit: participants
Arm/Group | Recombinant Human Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 30
participants | 23

2. Primary Outcome: Number of Participants Who Had at Least One Follicle Greater Than 17mm in Diameter
Time Frame: Day 14
Population: Per protocol set included all participants who completely met all the requirements of clinical trial protocol.
Measure: Number; unit: participants
Arm/Group | Recombinant Human Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 30
participants | 23

3. Primary Outcome: Number of Participants With E2 Level in Blood Serum Above 109 pg/mL on the Day of hCG Injection
Time Frame: Day 14
Population: Per protocol set included all participants who completely met all the requirements of clinical trial protocol.
Measure: Number; unit: participants
Arm/Group | Recombinant Human Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 30
participants | 23

4. Primary Outcome: Number of Participants Who Refused to Take hCG Injection
Description: Participant refused to take hCG injection for the concern of OHSS or the participant was pregnant.
Time Frame: Day 14
Population: Per protocol set included all participants who completely met all the requirements of clinical trial protocol.
Measure: Number; unit: participants
Arm/Group | Recombinant Human Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 30
participants
  Refused due to concern of OHSS | 0
  Refused due to pregnancy | 10

5. Secondary Outcome: Mean Number of Follicles With Diameter in the Range of 10-17 mm on the Day of hCG Injection in Treatment Cycle
Time Frame: Day 14
Population: Per protocol set included all participants who completely met all the requirements of clinical trial protocol.
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | Recombinant Human Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 30
follicles | 3.57 (4.07)

6. Secondary Outcome: Mean Number of Follicles With the Diameter Above 17 mm on the Day of hCG Injection in Treatment Cycle
Time Frame: Day 14
Population: Per protocol set included all participants who completely met all the requirements of clinical trial protocol.
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | Recombinant Human Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 30
follicles | 2.13 (2.00)

7. Secondary Outcome: Average Change of E2 Level in Participants Per Day up to Day 14
Description: The average change was calculated by assessing the E2 levels on 4 timepoints until day 14 (day 1, day 5, day 10, day 14 [hCG administration day]).
Time Frame: up to Day 14
Population: Per protocol set included all participants who completely met all the requirements of clinical trial protocol.
Measure: Mean (Standard Deviation); unit: pg/mL per day
Arm/Group | Recombinant Human Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 30
pg/mL per day | 71.03 (64.53)

8. Secondary Outcome: Number of Participants With Confirmed Pregnancies: Biochemical Pregnancies and Clinical Pregnancies
Description: Biochemical pregnancy was defined as a pregnancy diagnosed only by the detection of hCG in serum or urine and that does not develop into a clinical pregnancy. Clinical pregnancy was defined as a pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy. It includes ectopic pregnancy.
Time Frame: Day 14
Population: Per protocol set included all participants who completely met all the requirements of clinical trial protocol.
Measure: Number; unit: participants
Arm/Group | Recombinant Human Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 30
participants
  Biochemical Pregnancies | 1
  Clinical Pregnancies | 9

9. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any new untoward medical occurrence/worsening of pre-existing medical condition, whether or not related to study drug. SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was a medically important condition.
Time Frame: Day 14
Population: Safety analysis set included all participants who received investigational drug for at least one time.
Measure: Number; unit: participants
Arm/Group | Recombinant Human Luteinizing Hormone (Luveris)
Number analyzed (Participants) | 31
participants
  Adverse Events | 0
  Serious Adverse Events | 0

ADVERSE EVENTS:
Time Frame: Day 14
Description: An AE was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Recombinant Human Luteinizing Hormone (Luveris)
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other